CLINICAL TRIAL: NCT07379866
Title: Ultrasound Guided Glossopharyngeal and Maxillary Nerve Blocks for Perioperative Pain Control in Adenotonsillectomy in Pediatrics: A Randomized Controlled Trial.
Brief Title: Glossopharyngeal and Maxillary Nerve Blocks in Adenotonsillectomy
Acronym: Pediatrics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nagy Malak , MD, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS-389-2025; University (Other: Cairo University)
Record Dates: First submitted 2025-11-24; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Regional; Adenotonsillectomy
Keywords: Ultrasound; Glossopharyngeal; Adenotonsillectomy; Pediatrics

STUDY DESIGN:
Intervention Model Description: Patients will receive combined bilateral ultrasound-guided glossopharyngeal nerve (UGGNB) and bilateral ultrasound-guided maxillary nerve (UGMNB) immediately after the induction of anesthesia and prior to surgical incision by an expert anesthesiologist in ultrasound guided regional anesthesia who is not a part of the study using Philips Model HD5 Diagnostic ultrasound system a the scanning probe will be the linear ultrasound probe (4-12MHz) for glossopharyngeal nerve block and a curvilinear ultrasound probe (5-7 MHz) for maxillary nerve block using fine needle as described with aid of ultrasound.
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomization will be achieved using a computer-generated sequence. Concealment will be achieved using opaque envelopes. The study will be a single blinded trial where the assessor who follow the patients post-operatively is blinded to the technique given.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Block Group (Active Comparator): patients will receive combined bilateral ultrasound-guided glossopharyngeal nerve (UGGNB) and bilateral ultrasound-guided maxillary nerve (UGMNB) immediately after the induction of anesthesia and prior to surgical incision
  Interventions: Procedure: ultrasound-guided glossopharyngeal nerve block (UGSGNB); Procedure: ultrasound-guided maxillary nerve (UGMN)
- Conventional Group (Placebo Comparator): patients will receive multimodal analgesia for tonsillectomy operations in the form of single dose of IV paracetamol 15 mg/kg
  Interventions: Procedure: Placebo Block

INTERVENTIONS:
Procedure: ultrasound-guided glossopharyngeal nerve block (UGSGNB) — For the procedure, anesthesiologist will turn patient face carefully toward the clinician, and a linear ultrasound probe will be placed in the neck to check the surrounding target structures: the sternocleidomastoid muscle, the common carotid artery, and the internal jugular vein. After the sternocleidomastoid muscle has been identified, a linear ultrasound probe will be placed parallel to sternocleidomastoid muscle fiber direction just caudal to the mandibular ramus. The stylohyoid muscle is easily visualized by tiling the linear ultrasound probe toward the mandibular ramus. In this area, the stylohyoid muscle is positioned under the sternocleidomastoid muscle, and both can be observed under ultrasound guidance. A 25-gauge, 25-mm needle will be inserted deeply under the stylohyoid muscle through the sternocleidomastoid muscle via an out-of-plane approach. An ultrasound-guided nerve block will be performed with 3 mL of 0.25% bupivacaine after the absence of blood backflow is confirmed.
  Arms: Block Group
Procedure: ultrasound-guided maxillary nerve (UGMN) — Curvilinear ultrasound probe will be placed in infra-zygomatic area, over maxilla, angled 45° cephalad. This probe position allows visualization of pterygopalatine fossa, limited anteriorly by maxilla and posteriorly by greater wing of sphenoid. A 22- gauge, 5-cm needle will be inserted perpendicularly to the skin following aseptic preparation of the skin at the frontozygomatic angle formed by posterior orbital rim and zygomatic. Once contact was made with the greater wing of sphenoid, needle will be redirected caudally and medially, and advances through the pterygomaxillary fissure into pterygomaxillary fossa. needle will be advanced using an out-of-plane approach, and needle tip can usually be identified during movements.
  Needle placement will be verified by real-time ultrasound guidance and negative aspiration before administration of 3-4 ml of 0.25 % bupivacaine. The same procedure will be then repeated on the contralateral side.
  Arms: Block Group
Procedure: Placebo Block — ultrasound-guided maxillary nerve (UGMN) and ultrasound-guided glossopharyngeal nerve block (UGSGNB) using normal saline as placebo effect
  Arms: Conventional Group

SUMMARY:
This study aims to compare of bilateral ultrasound-guided glossopharyngeal nerve (UGGNB) and ultrasound-guided maxillary nerve (UGMNB) versus conventional multimodal analgesia for tonsillectomy operations.

DETAILED DESCRIPTION:
Patients will be premedicated with oral midazolam 0.5 mg/kg prior to arriving in the operating room 30 min before the procedure.

Standard monitoring will be maintained throughout the procedure included electrocardiography, noninvasive arterial pressure, arterial oxygen saturation.

. If intravenous access is present, Fentanyl 1 μg/kg IV will be given and anesthesia will be induced using propofol 2-3 mg/kg and atracurium 0.5 mg/kg. If intravenous access is not present, anesthesia will be induced with inhalation of 8% sevoflurane in 100% oxygen under spontaneous ventilation and IV access will be established, fentanyl 1 µg/kg IV and atracurium 0.5 m g/kg IV will be given after achieving IV access. Endotracheal intubation will be done using an appropriate size endotracheal tube (ETT) and capnography attached. IV dexamethasone 150 μg/kg will be given. Anesthesia will be maintained using a 50:50 mixture of air and oxygen along with isoflurane 1.2% and the maintenance dose of atracurium 0.1 mg/kg each 20 minutes. Pressure-controlled ventilation and low fresh gas flows will be used. All patients will receive intraoperative analgesia in the form of single dose paracetamol 15 mg/kg.

Patients will be randomly allocated into two equal groups:

Block Group: patients will receive combined bilateral ultrasound-guided glossopharyngeal nerve (UGGNB) and bilateral ultrasound-guided maxillary nerve (UGMNB) immediately after the induction of anesthesia and prior to surgical incision by an expert anesthesiologist in ultrasound guided regional anesthesia who is not a part of the study using Philips Model HD5 Diagnostic ultrasound system a the scanning probe will be the linear ultrasound probe (4-12MHz) for glossopharyngeal nerve block and a curvilinear ultrasound probe (5-7 MHz) for maxillary nerve block using fine needle as described with aid of ultrasound.

Conventional Group: patients will receive multimodal analgesia for tonsillectomy operations in the form of single dose of IV paracetamol 15 mg/kg.

Tonsillectomies will be carried out by expert surgeon using the same electro-dissection surgical technique.

In block group:

Technique of ultrasound-guided glossopharyngeal nerve block (UGSGNB): posterior mandibular ramus approach For the procedure, anesthesiologist will turn patient face carefully toward the clinician, and a linear ultrasound probe will be placed in the neck to check the surrounding target structures: the sternocleidomastoid muscle, the common carotid artery, and the internal jugular vein. After the sternocleidomastoid muscle has been identified, a linear ultrasound probe will be placed parallel to the sternocleidomastoid muscle fiber direction just caudal to the mandibular ramus. The stylohyoid muscle is easily visualized by tiling the linear ultrasound probe toward the mandibular ramus. In this area, the stylohyoid muscle is positioned under the sternocleidomastoid muscle, and both can be observed under ultrasound guidance. A 25-gauge, 25-mm needle will be inserted deeply under the stylohyoid muscle through the sternocleidomastoid muscle via an out-of-plane approach. An ultrasound-guided nerve block will be performed with 3 mL of 0.25% bupivacaine after the absence of blood backflow is confirmed. The same procedure will be then repeated on the contralateral side.

Technique of ultrasound-guided maxillary nerve (UGMNB): Suprazygomatic maxillary nerve blocks The curvilinear ultrasound probe will be placed in the infrazygomatic area, over the maxilla, angled 45° cephalad. This probe position allows visualization of the pterygopalatine fossa, limited anteriorly by the maxilla and posteriorly by the greater wing of the sphenoid. A 22- gauge, 5-cm nerve block needle will be inserted perpendicularly to the skin following aseptic preparation of the skin at the frontozygomatic angle formed by the posterior orbital rim and zygomatic . Once contact was made with the greater wing of the sphenoid, the needle will be redirected caudally and medially, and advances through the pterygomaxillary fissure into the pterygomaxillary fossa. The needle will be advanced using an out-of-plane approach, and the needle tip can usually be identified during movements.

Needle placement will be verified by real-time ultrasound guidance and negative aspiration before administration of 3-4 ml of 0.25 % bupivacaine. The same procedure will be then repeated on the contralateral side.

In both groups Baseline hemodynamics in the form of: non-invasive BP, HR, oxygen saturation will be recorded before induction of anesthesia. the intraoperative hemodynamics will be recorded at 15 minute intervals in addition to continuous monitoring of HR and oxygen saturation. If heart rate (HR) increases more than 20% of baseline an additional dose of fentanyl 1 µg/kg will be given , if blood pressure exceeding 20% from baseline an additional dose of fentanyl 1 µg/kg will be given with a maximum total dose of 5 mcg/kg if additional doses are required , if bradycardic atropine 0.01 mg/kg will be given. At the end of the surgery , Inhalational anesthesia will be discontinued and muscle relaxation will be reversed by atropine (0.02 mg/Kg) and neostigmine (0.05 mg/Kg) after the restoration of the patient's spontaneous breathing. The patient will be transferred to the post-anesthesia care unit (PACU) for 1 hours to complete recovery and monitoring and then will be sent to the ward. Quality of analgesia will be assessed using the Wong-Baker FACES scale for children more than 3 years of age up to 8 years of age and VAS score for older children every 30 minutes for 1 hours after recovery from anesthesia in PACU and every 2, 4, 8, 12, and 24 hours postoperative after transferring to the ward.

For postoperative pain therapy, If the pain scale scores are ≥ 4, first will be IV ibuprofen 7.5 mg/kg immediately postoperative.

Regarding that maximum single dose of ibuprofen is 400mg , maximum daily dose is 40mg/kg .

Paracetamol will not be given within 6 hour of intraoperative administration. After 15 mins if the pain scale scores still ≥ 4, patients will receive pethidine 0.5 mg/kg I.V. as rescue analgesia, which may be repeated, taking in consideration that the total daily dose should not exceed 1.5 mg/kg(11), regarding that minimum period of pethidine rescue analgesic doses are from 2 to 4 hours and. The analgesic effect occurs after about 10 minutes following parenteral administration.

Antiemetics (IV 1.25 mg/kg dimenhydrinate or 0.15 mg/kg of metoclopramide or 0.1 mg/kg ondansetron) will be given in the case of postoperative nausea and vomiting .

The patient will be discharged when the pain is controlled as the pain scale < 3 and there is no nausea, vomiting, and/or bleeding. Post discharge, the FACES and VAS scales will be explained to the parents for further assessment of pain score post-operative day for 24 hrs.

The parents will be contacted by phone numbers to asses pain score and the dose of paracetamol & ibuprofen will be documented.

Possible complications of local anesthetic toxicity will appear as hemodynamic instability in the form of hypotension and bradycardia and will be managed using bolus of crystalloids (20ml/kg),ephedrine (1-3mg) boluses and atropine (0.01mg/kg).

Any complications resulting from peripheral nerve blockade like: bleeding, infection or neuropathy, will be recorded and managed accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 5 to 13 years
* American Society of Anesthesiologists (ASA) physical status I-II scheduled for adenotonsillectomy.

Exclusion Criteria:

* Parents Refusal
* Cognitive impairment or developmental delays.
* Infection at injection site.
* Recent upper respiratory tract infection.
* Post-tonsillectomy bleeding, allergy to local anesthetics.
* American Society of Anesthesiologists (ASA) class III and IV.
* Morbid obesity.
* Those receiving regular analgesia within the last week before surgery.

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Time to first rescue analgesia | 24 hours
  Time of the first claim for analgesia

SECONDARY OUTCOMES:
Heart rate | 2 hours
  Intraoperative monitoring of heart rate measured beats/minute
Intraoperative fentanyl consumption | 2 hours
  Intraoperative fentanyl consumption in microgram
Dietary intake | 24 hours
  Dietary intake on post operative day 1 will be evaluated on a 5-point Likert scale (0 = no food intake; 5 = complete meals) at each meal by the ward nurse
Postoperative pain scores | 24 hours
  Postoperative pain scores every 2, 4, 8, 12, and 24 hours postoperative after transferring to the ward.
  Quality of analgesia will be assessed using Wong-Baker FACES scale for children more than 3 years of age up to 8 years of age and Visual Analogue Scale for older children every 30 minutes for 1 hour after recovery from anesthesia in PACU and every 2, 4, 8, 12, and 24 hours postoperative after transferring to ward.
Total pethidine requirements | 24 hours
  Total pethidine requirements 24 hours postoperatively.
Post tonsillectomy bleeding. | 24 hours
  Post tonsillectomy bleeding.
Blood Pressure | 2 hours
  intraoperative monitoring of Systolic, diastolic and Mean Blood Pressure mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Nagy malak, MD, Principal Investigator — Cairo University
Locations (1):
- Cairo University Hospitals, Cairo, Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No